CLINICAL TRIAL: NCT04279574
Title: Clinical Performance of Chairside CAD/CAM Restorations Using a New Adhesive Cement
Brief Title: Clinical Performance of Chairside CAD/CAM Restorations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Solventum US LLC (Industry)
Collaborators: University of Michigan (Other); 3M (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EM-11-050060
Record Dates: First submitted 2020-02-13; First posted 2020-02-21 (Actual); Results first posted 2025-03-24 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Dental Cements; Caries,Dental
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- CAD/CAM Onlays (Other): Lithium disilicate chairside CAD/CAM onlays (IPS emaxCAD/Ivoclar) will be adhesively bonded using a selective enamel etch technique with an adhesive (3M) and cement (3M).
  Interventions: Device: Lithium disilicate onlays (IPS emaxCAD/Ivoclar)
- CAD/CAM Crowns (Other): Full contour zirconia crowns (3M Chairside Zirconia/3M) will be cemented using a self-adhesive cement (3M).
  Interventions: Device: Chairside zirconia crowns (3M)

INTERVENTIONS:
Device: Lithium disilicate onlays (IPS emaxCAD/Ivoclar) — Restoration of posterior teeth
  Arms: CAD/CAM Onlays
Device: Chairside zirconia crowns (3M) — Restoration of posterior teeth
  Arms: CAD/CAM Crowns

SUMMARY:
This investigation will be a longitudinal clinical trial to study the long-term clinical performance of a resin cement for chairside CAD/CAM restorations. Lithium disilicate chairside CAD/CAM onlays will be adhesively bonded using a selective enamel etch technique with an adhesive.

Full contour zirconia crowns will be cemented using a self-adhesive resin cement.

DETAILED DESCRIPTION:
A wide variety of restorative materials are available for dental restorations. The most popular current materials include glass ceramics and full contour zirconia. Glass ceramic materials are generally preferred for their high translucency mimicking enamel-like esthetics of natural teeth and zirconia is preferred for high strength applications. Both of these materials are available for clinical treatment using chairside CAD/CAM technology.

The introduction of an induction sintering oven (SpeedFire oven/Dentsply Sirona) opened the opportunity for chairside full contour zirconia crowns by decreasing sintering times for zirconia to under 30 minutes. 3M Chairside Zirconia (3M) was marketed in 2019 and offers improved esthetics and high strength for monolithic zirconia restorations with an efficient processing time.

This investigation will be a longitudinal clinical trial to study the long-term clinical performance of CAD/CAM restorations. Lithium disilicate chairside CAD/CAM onlays (IPS emaxCAD/Ivoclar) will be adhesively bonded using a selective enamel etch technique with a universal adhesive (3M) and a resin cement (3M). Full contour zirconia crowns (3M Chairside Zirconia/3M) will be cemented using a self-adhesive technique.

ELIGIBILITY:
Inclusion Criteria:

* Subject in need of crown and/or onlay restoration
* Subject age 18 or above
* Subject with healthy / treated periodontal status (max. degree of movement 1)
* Subject agrees to participate in the study and signed informed consent and HIPAA form

Exclusion Criteria:

* Devital or sensitive teeth
* Teeth diagnosed with symptoms of incomplete tooth fracture
* Teeth with prior endodontic treatment of any kind
* Teeth with a history of direct or indirect pulp capping procedures
* Subjects with uncontrolled bruxism or parafunctional habits
* Subject has known allergies to any product used in this study
* Subject will not be available for the study duration
* Subjects with significant untreated dental disease to include periodontitis and rampant caries
* Pregnant or lactating women

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2020-08-26 (Actual); Primary Completion 2024-05-22 (Actual); Study Completion 2024-05-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paula Myhre, Study Director — Solventum
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hickel R, Peschke A, Tyas M, Mjor I, Bayne S, Peters M, Hiller KA, Randall R, Vanherle G, Heintze SD. FDI World Dental Federation: clinical criteria for the evaluation of direct and indirect restorations-update and clinical examples. Clin Oral Investig. 2010 Aug;14(4):349-66. doi: 10.1007/s00784-010-0432-8. Epub 2010 Jul 14. PMID 20628774
- [Background] SILNESS J, LOE H. PERIODONTAL DISEASE IN PREGNANCY. II. CORRELATION BETWEEN ORAL HYGIENE AND PERIODONTAL CONDTION. Acta Odontol Scand. 1964 Feb;22:121-35. doi: 10.3109/00016356408993968. No abstract available. PMID 14158464
- [Background] LOE H, SILNESS J. PERIODONTAL DISEASE IN PREGNANCY. I. PREVALENCE AND SEVERITY. Acta Odontol Scand. 1963 Dec;21:533-51. doi: 10.3109/00016356309011240. No abstract available. PMID 14121956

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The patient population was selected from current patients under clinical treatment at the University of Michigan Dental Clinics. Patients were over 18 years of age, of either gender, and of any ethnic background. Each patient had at least one carious lesion or defective restoration to be restored on a maxillary or mandibular premolar or molar tooth.
Pre-assignment Details: Each lesion or defective restoration exhibited sufficient size to extend at least one-half the intercuspal width of the tooth requiring an onlay or full crown restoration. The onlays covered between one and three cusps on the selected tooth and maintained an occlusal margin. All teeth tested vital and were asymptomatic at the beginning of treatment. No more than two restorations were placed per patient; molar teeth were included prior to premolar teeth.
Units Other Than Participants: Restorations
Period: Overall Study
Arm/Group | CAD/CAM Onlays | CAD/CAM Crowns
Started (Up to two restorations of either type (onlays and/or crowns) were allowed per subject. Actual overall number of participants treated was 58.) | 35; 40 Restorations | 33; 40 Restorations
Completed | 33; 38 Restorations | 32; 39 Restorations
Not Completed | 2; 2 Restorations | 1; 1 Restorations
Not completed — Death | 1 | 0
Not completed — lost restoration, tooth fracture | 1 | 0
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Population: Up to two restorations of either type (onlays and/or crowns) were allowed per subject. Actual overall number of participants treated was 58. Of the 58 subjects, 36 had one restoration and 22 had two restorations.
Units Other Than Participants: Number of Teeth Treated
Groups:
- Total: Total of all reporting groups
Arm/Group | CAD/CAM Onlays | CAD/CAM Crowns | Total
Number analyzed (Participants) | 35 | 33 | 58
Number analyzed (Number of Teeth Treated) | 40 | 40 | 80
Age, Continuous [Mean (Standard Deviation); unit: years] — Age at time of consent, subjects must be 18 years of age or older. Population: Up to two restorations of either type (onlays and/or crowns) were allowed per subject. Actual overall number of participants treated was 58.
  years | 59 (9) | 63 (8) | 61 (9)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Up to two restorations of either type (onlays and/or crowns) were allowed per subject. Actual overall number of participants treated was 58.
  Participants
    Female | 25 | 25 | 50
    Male | 10 | 8 | 18
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
  Participants
    number analyzed (Participants) | 0 | 0 | 0
    (all) |  |  | 0
Type of restoration [Count of Units; unit: Number of Teeth Treated] — Number of Onlays and Number of Crowns. Population: Up to two restorations of either type (onlays and/or crowns) were allowed per subject. Actual overall number of participants treated was 58.
  Number of Teeth Treated
    Premolars | 10 | 6 | 16
    Molars | 30 | 34 | 64

OUTCOME MEASURES:

1. Primary Outcome: Functional Long-term Properties Clinical Performance of Restorations (Onlays and Crowns) [Retention Scores]
Description: Retention. Evaluations according to FDI World Dental Federation criteria (Hickel et al., 2010) [5b.1 Restoration in place; 5b.5 Complete loss of restoration] Functional property (retention) assessed by visual and/or tactile assessment by two independent examiners.]
Time Frame: 3 years with assessment visits at baseline, 6 months, 1 year, 2 years, and 3 years
Population: Up to two restorations of either type (onlays and/or crowns) were allowed per subject. Actual overall number of participants treated was 58.
Measure: Count of Units; unit: Restorations
Units Other Than Participants: Restorations
Arm/Group | CAD/CAM Onlays | CAD/CAM Crowns
Number analyzed (Participants) | 35 | 33
Number analyzed (Restorations) | 40 | 40
Restorations
  Baseline: 5b.1 Restoration in place | 40 | 40
  Baseline: 5b.5 Complete loss of restoration | 0 | 0
  Baseline: Missed visit / no data | 0 | 0
  Baseline: Failed Onlay / Crown | 0 | 0
  6 months post-restoration: 5b.1 Restoration in place | 40 | 40
  6 months post-restoration: 5b.5 Complete loss of restoration | 0 | 0
  6 months post-restoration: Missed visit / no data | 0 | 0
  6 months post-restoration: Failed Onlay / Crown | 0 | 0
  1 year post-restoration: 5b.1 Restoration in place | 39 | 39
  1 year post-restoration: 5b.5 Complete loss of restoration | 0 | 0
  1 year post-restoration: Missed visit / no data | 1 | 1
  1 year post-restoration: Failed Onlay / Crown | 0 | 0
  2 years post-restoration: 5b.1 Restoration in place | 37 | 39
  2 years post-restoration: 5b.5 Complete loss of restoration | 2 | 1
  2 years post-restoration: Missed visit / no data | 0 | 0
  2 years post-restoration: Failed Onlay / Crown | 1 | 0
  3 years post-restoration: 5b.1 Restoration in place | 36 | 38
  3 years post-restoration: 5b.5 Complete loss of restoration | 2 | 1
  3 years post-restoration: Missed visit / no data | 1 | 1
  3 years post-restoration: Failed Onlay / Crown | 1 | 0

2. Secondary Outcome: Functional Long-term Properties Clinical Performance of Restorations (Onlays and Crowns) [Material Fracture Scores]
Description: Material Fracture. Evaluations according to FDI World Dental Federation criteria (Hickel et al., 2010) [1: Clinically excellent, 2: Clinically good, 3: Clinically sufficient, 4: Clinically unsatisfactory, 5: Clinically poor] Functional properties assessed by visual and/or tactile assessment by two independent examiners.]
Time Frame: 3 years with assessment visits at baseline, 6 months, 1 year, 2 years, and 3 years
Population: as for outcome 1
Measure: Count of Units; unit: Restorations
Units Other Than Participants: Restorations
Arm/Group | CAD/CAM Onlays | CAD/CAM Crowns
Number analyzed (Participants) | 35 | 33
Number analyzed (Restorations) | 40 | 40
Restorations
  Baseline: 1: Clinically excellent | 40 | 40
  Baseline: 2: Clinically good | 0 | 0
  Baseline: Missed visit / no data | 0 | 0
  Baseline: Failed Onlay / Crown | 0 | 0
  6 months post-restoration: 1: Clinically excellent | 40 | 40
  6 months post-restoration: 2: Clinically good | 0 | 0
  6 months post-restoration: Missed visit / no data | 0 | 0
  6 months post-restoration: Failed Onlay / Crown | 0 | 0
  1 year post-restoration: 1: Clinically excellent | 39 | 39
  1 year post-restoration: 2: Clinically good | 0 | 0
  1 year post-restoration: Missed visit / no data | 1 | 1
  1 year post-restoration: Failed Onlay / Crown | 0 | 0
  2 years post-restoration: 1: Clinically excellent | 39 | 40
  2 years post-restoration: 2: Clinically good | 0 | 0
  2 years post-restoration: Missed visit / no data | 0 | 0
  2 years post-restoration: Failed Onlay / Crown | 1 | 0
  3 years post-restoration: 1: Clinically excellent | 38 | 39
  3 years post-restoration: 2: Clinically good | 0 | 0
  3 years post-restoration: Missed visit / no data | 1 | 1
  3 years post-restoration: Failed Onlay / Crown | 1 | 0

3. Secondary Outcome: Functional Long-term Properties Clinical Performance of Restorations (Onlays and Crowns) [Approximal Anatomical Contact Form - Mesial]
Description: Approximal anatomical contact form - mesial. Evaluations according to FDI World Dental Federation criteria (Hickel et al., 2010) [1: Clinically excellent, 2: Clinically good, 3: Clinically sufficient, 4: Clinically unsatisfactory, 5: Clinically poor] Functional property assessed by visual and/or tactile assessment by two independent examiners.]
Time Frame: 3 years with assessment visits at baseline, 6 months, 1 year, 2 years, and 3 years
Population: as for outcome 1
Measure: Count of Units; unit: Restorations
Units Other Than Participants: Restorations
Arm/Group | CAD/CAM Onlays | CAD/CAM Crowns
Number analyzed (Participants) | 35 | 33
Number analyzed (Restorations) | 40 | 40
Restorations
  Baseline: 1: Clinically excellent | 38 | 40
  Baseline: 2: Clinically good | 0 | 0
  Baseline: Missed visit / no data | 0 | 0
  Baseline: Not applicable | 2 | 0
  Baseline: Failed onlay / crown | 0 | 0
  6 months post-restoration: 1: Clinically excellent | 36 | 40
  6 months post-restoration: 2: Clinically good | 0 | 0
  6 months post-restoration: Missed visit / no data | 0 | 0
  6 months post-restoration: Not applicable | 4 | 0
  6 months post-restoration: Failed onlay / crown | 0 | 0
  1 year post-restoration: 1: Clinically excellent | 34 | 39
  1 year post-restoration: 2: Clinically good | 0 | 0
  1 year post-restoration: Missed visit / no data | 1 | 1
  1 year post-restoration: Not applicable | 5 | 0
  1 year post-restoration: Failed onlay / crown | 0 | 0
  2 years post-restoration: 1: Clinically excellent | 34 | 40
  2 years post-restoration: 2: Clinically good | 0 | 0
  2 years post-restoration: Missed visit / no data | 0 | 0
  2 years post-restoration: Not applicable | 5 | 0
  2 years post-restoration: Failed onlay / crown | 1 | 0
  3 years post-restoration: 1: Clinically excellent | 33 | 39
  3 years post-restoration: 2: Clinically good | 0 | 0
  3 years post-restoration: Missed visit / no data | 1 | 1
  3 years post-restoration: Not applicable | 5 | 0
  3 years post-restoration: Failed onlay / crown | 1 | 0

4. Secondary Outcome: Functional Long-term Properties Clinical Performance of Restorations (Onlays and Crowns) [Approximal Anatomical Contact Point - Mesial Scores]
Description: Approximal anatomical contact point - mesial. Evaluations according to FDI World Dental Federation criteria (Hickel et al., 2010) [1: Clinically excellent, 2: Clinically good, 3: Clinically sufficient, 4: Clinically unsatisfactory, 5: Clinically poor] Functional property assessed by visual and/or tactile assessment by two independent examiners.]
Time Frame: 3 years with assessment visits at baseline, 6 months, 1 year, 2 years, and 3 years
Population: as for outcome 1
Measure: Count of Units; unit: Restorations
Units Other Than Participants: Restorations
Arm/Group | CAD/CAM Onlays | CAD/CAM Crowns
Number analyzed (Participants) | 35 | 33
Number analyzed (Restorations) | 40 | 40
Restorations
  Baseline: 1: Clinically excellent | 38 | 40
  Baseline: 2: Clinically good | 0 | 0
  Baseline: 3: Clinically sufficient | 0 | 0
  Baseline: Missed visit / no data | 0 | 0
  Baseline: Failed Onlay / Crown | 0 | 0
  Baseline: Not Applicable | 2 | 0
  6 months post-restoration: 1: Clinically excellent | 35 | 39
  6 months post-restoration: 2: Clinically good | 0 | 0
  6 months post-restoration: 3: Clinically sufficient | 1 | 1
  6 months post-restoration: Missed visit / no data | 0 | 0
  6 months post-restoration: Failed Onlay / Crown | 0 | 0
  6 months post-restoration: Not Applicable | 4 | 0
  1 year post-restoration: 1: Clinically excellent | 33 | 37
  1 year post-restoration: 2: Clinically good | 0 | 0
  1 year post-restoration: 3: Clinically sufficient | 1 | 2
  1 year post-restoration: Missed visit / no data | 1 | 1
  1 year post-restoration: Failed Onlay / Crown | 0 | 0
  1 year post-restoration: Not Applicable | 5 | 0
  2 years post-restoration: 1: Clinically excellent | 34 | 39
  2 years post-restoration: 2: Clinically good | 0 | 0
  2 years post-restoration: 3: Clinically sufficient | 0 | 1
  2 years post-restoration: Missed visit / no data | 0 | 0
  2 years post-restoration: Failed Onlay / Crown | 1 | 0
  2 years post-restoration: Not Applicable | 5 | 0
  3 years post-restoration: 1: Clinically excellent | 33 | 39
  3 years post-restoration: 2: Clinically good | 0 | 0
  3 years post-restoration: 3: Clinically sufficient | 0 | 0
  3 years post-restoration: Missed visit / no data | 1 | 1
  3 years post-restoration: Failed Onlay / Crown | 1 | 0
  3 years post-restoration: Not Applicable | 5 | 0

5. Secondary Outcome: Functional Long-term Properties Clinical Performance of Restorations (Onlays and Crowns) [Approximal Anatomical Contact Form - Distal Scores]
Description: Approximal Anatomical Contact Form - Distal. Evaluations according to FDI World Dental Federation criteria (Hickel et al., 2010) [1: Clinically excellent, 2: Clinically good, 3: Clinically sufficient, 4: Clinically unsatisfactory, 5: Clinically poor] Functional property assessed by visual and/or tactile assessment by two independent examiners.]
Time Frame: 3 years with assessment visits at baseline, 6 months, 1 year, 2 years, and 3 years
Population: as for outcome 1
Measure: Count of Units; unit: Restorations
Units Other Than Participants: Restorations
Arm/Group | CAD/CAM Onlays | CAD/CAM Crowns
Number analyzed (Participants) | 35 | 33
Number analyzed (Restorations) | 40 | 40
Restorations
  Baseline: 1: Clinically excellent | 29 | 25
  Baseline: 2: Clinically good | 0 | 0
  Baseline: Missed visit / no data | 0 | 0
  Baseline: Failed Onlay / Crown | 0 | 0
  Baseline: Not Applicable | 11 | 15
  6 months post-restoration: 1: Clinically excellent | 27 | 24
  6 months post-restoration: 2: Clinically good | 0 | 0
  6 months post-restoration: Missed visit / no data | 0 | 0
  6 months post-restoration: Failed Onlay / Crown | 0 | 0
  6 months post-restoration: Not Applicable | 13 | 16
  1 year post-restoration: 1: Clinically excellent | 27 | 22
  1 year post-restoration: 2: Clinically good | 0 | 0
  1 year post-restoration: Missed visit / no data | 1 | 1
  1 year post-restoration: Failed Onlay / Crown | 0 | 0
  1 year post-restoration: Not Applicable | 12 | 17
  2 years post-restoration: 1: Clinically excellent | 26 | 24
  2 years post-restoration: 2: Clinically good | 0 | 0
  2 years post-restoration: Missed visit / no data | 0 | 0
  2 years post-restoration: Failed Onlay / Crown | 1 | 0
  2 years post-restoration: Not Applicable | 13 | 16
  3 years post-restoration: 1: Clinically excellent | 24 | 22
  3 years post-restoration: 2: Clinically good | 0 | 0
  3 years post-restoration: Missed visit / no data | 1 | 1
  3 years post-restoration: Failed Onlay / Crown | 1 | 0
  3 years post-restoration: Not Applicable | 14 | 17

6. Secondary Outcome: Functional Long-term Properties Clinical Performance of Restorations (Onlays and Crowns) [Approximal Anatomical Contact Point - Distal Scores]
Description: Approximal Anatomical Contact Point - Distal. Evaluations according to FDI World Dental Federation criteria (Hickel et al., 2010) [1: Clinically excellent, 2: Clinically good, 3: Clinically sufficient, 4: Clinically unsatisfactory, 5: Clinically poor] Functional property assessed by visual and/or tactile assessment by two independent examiners.]
Time Frame: 3 years with assessment visits at baseline, 6 months, 1 year, 2 years, and 3 years
Population: as for outcome 1
Measure: Count of Units; unit: Restorations
Units Other Than Participants: Restorations
Arm/Group | CAD/CAM Onlays | CAD/CAM Crowns
Number analyzed (Participants) | 35 | 33
Number analyzed (Restorations) | 40 | 40
Restorations
  Baseline: 1: Clinically excellent | 29 | 25
  Baseline: 2: Clinically good | 0 | 0
  Baseline: 3: Clinically sufficient | 0 | 0
  Baseline: Missed visit / no data | 0 | 0
  Baseline: Failed Onlay / Crown | 0 | 0
  Baseline: Not Applicabl | 11 | 15
  6 months post-restoration: 1: Clinically excellent | 27 | 24
  6 months post-restoration: 2: Clinically good | 0 | 0
  6 months post-restoration: 3: Clinically sufficient | 0 | 0
  6 months post-restoration: Missed visit / no data | 0 | 0
  6 months post-restoration: Failed Onlay / Crown | 0 | 0
  6 months post-restoration: Not Applicabl | 13 | 16
  1 year post-restoration: 1: Clinically excellent | 27 | 22
  1 year post-restoration: 2: Clinically good | 0 | 0
  1 year post-restoration: 3: Clinically sufficient | 0 | 0
  1 year post-restoration: Missed visit / no data | 1 | 1
  1 year post-restoration: Failed Onlay / Crown | 0 | 0
  1 year post-restoration: Not Applicabl | 12 | 17
  2 years post-restoration: 1: Clinically excellent | 26 | 23
  2 years post-restoration: 2: Clinically good | 0 | 0
  2 years post-restoration: 3: Clinically sufficient | 0 | 1
  2 years post-restoration: Missed visit / no data | 0 | 0
  2 years post-restoration: Failed Onlay / Crown | 1 | 0
  2 years post-restoration: Not Applicabl | 13 | 16
  3 years post-restoration: 1: Clinically excellent | 24 | 21
  3 years post-restoration: 2: Clinically good | 0 | 0
  3 years post-restoration: 3: Clinically sufficient | 0 | 1
  3 years post-restoration: Missed visit / no data | 1 | 1
  3 years post-restoration: Failed Onlay / Crown | 1 | 0
  3 years post-restoration: Not Applicabl | 14 | 17

7. Secondary Outcome: Functional Long-term Properties Clinical Performance of Restorations (Onlays and Crowns) [Occlusal Contour and Wear Scores]
Description: Occlusal contour and wear. Evaluations according to FDI World Dental Federation critera (Hickel et al., 2010) [1: Clinically excellent, 2: Clinically good, 3: Clinically sufficient, 4: Clinically unsatisfactory, 5: Clinically poor] Functional property assessed by visual and/or tactile assessment by two independent examiners.]
Time Frame: 3 years with assessment visits at baseline, 6 months, 1 year, 2 years, and 3 years
Population: as for outcome 1
Measure: Count of Units; unit: Restorations
Units Other Than Participants: Restorations
Arm/Group | CAD/CAM Onlays | CAD/CAM Crowns
Number analyzed (Participants) | 35 | 33
Number analyzed (Restorations) | 40 | 40
Restorations
  Baseline: 1: Clinically excellent | 40 | 40
  Baseline: 2: Clinically good | 0 | 0
  Baseline: Missed visit / no data | 0 | 0
  Baseline: Failed onlay / crown | 0 | 0
  6 months post-restoration: 1: Clinically excellent | 40 | 40
  6 months post-restoration: 2: Clinically good | 0 | 0
  6 months post-restoration: Missed visit / no data | 0 | 0
  6 months post-restoration: Failed onlay / crown | 0 | 0
  1 year post-restoration: 1: Clinically excellent | 39 | 39
  1 year post-restoration: 2: Clinically good | 0 | 0
  1 year post-restoration: Missed visit / no data | 1 | 1
  1 year post-restoration: Failed onlay / crown | 0 | 0
  2 years post-restoration: 1: Clinically excellent | 39 | 40
  2 years post-restoration: 2: Clinically good | 0 | 0
  2 years post-restoration: Missed visit / no data | 0 | 0
  2 years post-restoration: Failed onlay / crown | 1 | 0
  3 years post-restoration: 1: Clinically excellent | 38 | 37
  3 years post-restoration: 2: Clinically good | 0 | 2
  3 years post-restoration: Missed visit / no data | 1 | 1
  3 years post-restoration: Failed onlay / crown | 1 | 0

8. Secondary Outcome: Biologic Properties of Restorations (Onlays and Crowns) [Recurrence of Caries, Erosion, Abfraction Scores]
Description: Recurrence of caries, erosion, abfraction. Evaluations according to FDI World Dental Federation criteria (Hickel et al., 2010) [1: Clinically excellent, 2: Clinically good, 3: Clinically sufficient, 4: Clinically unsatisfactory, 5: Clinically poor] Biological properties assessed by visual and/or tactile assessment by two independent examiners.]
Time Frame: 3 years with assessments at 6 months, 1 year, 2 years, and 3 years
Population: as for outcome 1
Measure: Count of Units; unit: Restorations
Units Other Than Participants: Restorations
Arm/Group | CAD/CAM Onlays | CAD/CAM Crowns
Number analyzed (Participants) | 35 | 33
Number analyzed (Restorations) | 40 | 40
Restorations
  6 months post-restoration: 1: Clinically excellent | 40 | 40
  6 months post-restoration: 2: Clinically good | 0 | 0
  6 months post-restoration: 3: Clinically sufficient | 0 | 0
  6 months post-restoration: 4: Clinically unsatisfactory | 0 | 0
  6 months post-restoration: 5: Clinically poor | 0 | 0
  6 months post-restoration: Missed visit / no data | 0 | 0
  6 months post-restoration: Failed onlay / crown | 0 | 0
  1 year post-restoration: 1: Clinically excellent | 39 | 39
  1 year post-restoration: 2: Clinically good | 0 | 0
  1 year post-restoration: 3: Clinically sufficient | 0 | 0
  1 year post-restoration: 4: Clinically unsatisfactory | 0 | 0
  1 year post-restoration: 5: Clinically poor | 0 | 0
  1 year post-restoration: Missed visit / no data | 1 | 1
  1 year post-restoration: Failed onlay / crown | 0 | 0
  2 years post-restoration: 1: Clinically excellent | 39 | 40
  2 years post-restoration: 2: Clinically good | 0 | 0
  2 years post-restoration: 3: Clinically sufficient | 0 | 0
  2 years post-restoration: 4: Clinically unsatisfactory | 0 | 0
  2 years post-restoration: 5: Clinically poor | 0 | 0
  2 years post-restoration: Missed visit / no data | 0 | 0
  2 years post-restoration: Failed onlay / crown | 1 | 0
  3 years post-restoration: 1: Clinically excellent | 37 | 39
  3 years post-restoration: 2: Clinically good | 0 | 0
  3 years post-restoration: 3: Clinically sufficient | 0 | 0
  3 years post-restoration: 4: Clinically unsatisfactory | 0 | 0
  3 years post-restoration: 5: Clinically poor | 1 | 0
  3 years post-restoration: Missed visit / no data | 1 | 1
  3 years post-restoration: Failed onlay / crown | 1 | 0

9. Secondary Outcome: Functional Long-term Properties Clinical Performance of Restorations (Onlays and Crowns) [Marginal Adaptation Scores]
Description: Marginal Adaptation. Evaluations according to FDI World Dental Federation criteria (Hickel et al., 2010) [1: Clinically excellent, 2: Clinically good, 3: Clinically sufficient, 4: Clinically unsatisfactory, 5: Clinically poor] Functional property assessed by visual and/or tactile assessment by two independent examiners.]
Time Frame: 3 years with assessment visits at baseline, 6 months, 1 year, 2 years, and 3 years
Population: as for outcome 1
Measure: Count of Units; unit: Restorations
Units Other Than Participants: Restorations
Arm/Group | CAD/CAM Onlays | CAD/CAM Crowns
Number analyzed (Participants) | 35 | 33
Number analyzed (Restorations) | 40 | 40
Restorations
  Baseline: 1: Clinically excellent | 40 | 40
  Baseline: 2: Clinically good | 0 | 0
  Baseline: Missed visit / no data | 0 | 0
  Baseline: Failed onlay / crown | 0 | 0
  6 months post-restoration: 1: Clinically excellent | 31 | 31
  6 months post-restoration: 2: Clinically good | 9 | 9
  6 months post-restoration: Missed visit / no data | 0 | 0
  6 months post-restoration: Failed onlay / crown | 0 | 0
  1 year post-restoration: 1: Clinically excellent | 20 | 14
  1 year post-restoration: 2: Clinically good | 19 | 25
  1 year post-restoration: Missed visit / no data | 1 | 1
  1 year post-restoration: Failed onlay / crown | 0 | 0
  2 years post-restoration: 1: Clinically excellent | 12 | 9
  2 years post-restoration: 2: Clinically good | 27 | 31
  2 years post-restoration: Missed visit / no data | 0 | 0
  2 years post-restoration: Failed onlay / crown | 1 | 0
  3 years post-restoration: 1: Clinically excellent | 1 | 11
  3 years post-restoration: 2: Clinically good | 37 | 28
  3 years post-restoration: Missed visit / no data | 1 | 1
  3 years post-restoration: Failed onlay / crown | 1 | 0

10. Secondary Outcome: Esthetic Properties of Restorations (Onlays and Crowns) [Surface Luster Scores]
Description: Surface Luster: Evaluations according to FDI World Dental Federation criteria (Hickel et al., 2010) [1: Clinically excellent, 2: Clinically good, 3: Clinically sufficient, 4: Clinically unsatisfactory, 5: Clinically poor]
Time Frame: 3 years with assessment visits at baseline, 6 months, 1 year, 2 years, and 3 years
Population: as for outcome 1
Measure: Count of Units; unit: Restorations
Units Other Than Participants: Restorations
Arm/Group | CAD/CAM Onlays | CAD/CAM Crowns
Number analyzed (Participants) | 35 | 33
Number analyzed (Restorations) | 40 | 40
Restorations
  Baseline: 1: Clinically excellent | 40 | 40
  Baseline: 2: Clinically good | 0 | 0
  Baseline: Missed visit / no data | 0 | 0
  Baseline: Failed onlay / crown | 0 | 0
  6 months post-restoration: 1: Clinically excellent | 40 | 40
  6 months post-restoration: 2: Clinically good | 0 | 0
  6 months post-restoration: Missed visit / no data | 0 | 0
  6 months post-restoration: Failed onlay / crown | 0 | 0
  1 year post-restoration: 1: Clinically excellent | 39 | 39
  1 year post-restoration: 2: Clinically good | 0 | 0
  1 year post-restoration: Missed visit / no data | 1 | 1
  1 year post-restoration: Failed onlay / crown | 0 | 0
  2 years post-restoration: 1: Clinically excellent | 39 | 40
  2 years post-restoration: 2: Clinically good | 0 | 0
  2 years post-restoration: Missed visit / no data | 0 | 0
  2 years post-restoration: Failed onlay / crown | 1 | 0
  3 years post-restoration: 1: Clinically excellent | 38 | 39
  3 years post-restoration: 2: Clinically good | 0 | 0
  3 years post-restoration: Missed visit / no data | 1 | 1
  3 years post-restoration: Failed onlay / crown | 1 | 0

11. Secondary Outcome: Short-term Post-operative Sensitivity (Onlays and Crowns)
Description: Evaluations according to FDI World Dental Federation criteria (Hickel et al., 2010) [Rating Scale 1: Clinically excellent, 2: Clinically good, 3: Clinically sufficient, 4: Clinically unsatisfactory, 5: Clinically poor] Biological properties assessed by patient interview.
Time Frame: up to 4 weeks after baseline with weekly assessments or until the restoration is reported asymptomatic
Population: as for outcome 1
Measure: Count of Units; unit: Restorations
Units Other Than Participants: Restorations
Arm/Group | CAD/CAM Onlays | CAD/CAM Crowns
Number analyzed (Participants) | 35 | 33
Number analyzed (Restorations) | 40 | 40
Restorations
  1 week post-restoration: Clinically excellent | 37 | 34
  1 week post-restoration: Clinically good | 3 | 4
  1 week post-restoration: Clinically sufficient | 0 | 2
  1 week post-restoration: Not assessed | 0 | 0
  2 weeks post-restoration: Clinically excellent | 40 | 37
  2 weeks post-restoration: Clinically good | 0 | 2
  2 weeks post-restoration: Clinically sufficient | 0 | 1
  2 weeks post-restoration: Not assessed | 0 | 0
  3 weeks post-restoration: Clinically excellent | 0 | 40
  3 weeks post-restoration: Clinically good | 0 | 0
  3 weeks post-restoration: Clinically sufficient | 0 | 0
  3 weeks post-restoration: Not assessed | 40 | 0

12. Secondary Outcome: Gingival Index (Onlays and Crowns)
Description: Loe & Silness Index, 1963 [0: normal gingiva, 1: mild inflammation and no bleeding, 2: moderate inflammation and bleeding, 3: severe inflammation]
Time Frame: 3 years with assessments at 6 months, 1 year, 2 years, and 3 years
Population: as for outcome 1
Measure: Count of Units; unit: Restorations
Units Other Than Participants: Restorations
Arm/Group | CAD/CAM Onlays | CAD/CAM Crowns
Number analyzed (Participants) | 35 | 33
Number analyzed (Restorations) | 40 | 40
Restorations
  6 months post-restporation: 1. Normal gingiva | 40 | 40
  6 months post-restporation: 2: Moderate inflammation and bleeding | 0 | 0
  6 months post-restporation: Missed visit / no data | 0 | 0
  6 months post-restporation: Failed onlay / crown | 0 | 0
  1 year post-restoration: 1. Normal gingiva | 38 | 38
  1 year post-restoration: 2: Moderate inflammation and bleeding | 1 | 1
  1 year post-restoration: Missed visit / no data | 1 | 1
  1 year post-restoration: Failed onlay / crown | 0 | 0
  2 years post-restoration: 1. Normal gingiva | 39 | 39
  2 years post-restoration: 2: Moderate inflammation and bleeding | 0 | 1
  2 years post-restoration: Missed visit / no data | 0 | 0
  2 years post-restoration: Failed onlay / crown | 1 | 0
  3 years post-restoration: 1. Normal gingiva | 37 | 37
  3 years post-restoration: 2: Moderate inflammation and bleeding | 1 | 2
  3 years post-restoration: Missed visit / no data | 1 | 1
  3 years post-restoration: Failed onlay / crown | 1 | 0

13. Secondary Outcome: Plaque Index (Onlays and Crowns)
Description: Silness & Loe Index, 1964 [0: plaque detectable in the gingival area, 1: plaque recognized only by running tip of probe across tooth surface at gingival crest, 2: moderate accumulation of plaque visible along gingival margin and adjacent tooth, 3: abundance of plaque visible along gingival margin and adjacent tooth]
Time Frame: 3 years with assessments at 6 months, 1 year, 2 years, and 3 years
Population: as for outcome 1
Measure: Count of Units; unit: Restorations
Units Other Than Participants: Restorations
Arm/Group | CAD/CAM Onlays | CAD/CAM Crowns
Number analyzed (Participants) | 35 | 33
Number analyzed (Restorations) | 40 | 40
Restorations
  6 months post-retoration: 1: plaque recognized | 40 | 37
  6 months post-retoration: 2: moderate accumulation of plaque | 0 | 3
  6 months post-retoration: Missed visit / no data | 0 | 0
  6 months post-retoration: Failed onlay / crown | 0 | 0
  1 year post-restoration: 1: plaque recognized | 36 | 35
  1 year post-restoration: 2: moderate accumulation of plaque | 3 | 4
  1 year post-restoration: Missed visit / no data | 1 | 1
  1 year post-restoration: Failed onlay / crown | 0 | 0
  2 years post-restoration: 1: plaque recognized | 39 | 36
  2 years post-restoration: 2: moderate accumulation of plaque | 0 | 4
  2 years post-restoration: Missed visit / no data | 0 | 0
  2 years post-restoration: Failed onlay / crown | 1 | 0
  3 years post-restoration: 1: plaque recognized | 37 | 33
  3 years post-restoration: 2: moderate accumulation of plaque | 1 | 6
  3 years post-restoration: Missed visit / no data | 1 | 1
  3 years post-restoration: Failed onlay / crown | 1 | 0

14. Secondary Outcome: Esthetic Properties Clinical Performance of Restorations (Onlays and Crowns) [Aesthetic Anatomical Form]
Description: Aesthetic Anatomical Form. Evaluations according to FDI World Dental Federation criteria (Hickel et al., 2010) [1: Clinically excellent, 2: Clinically good, 3: Clinically sufficient, 4: Clinically unsatisfactory, 5: Clinically poor] Functional property assessed by visual and/or tactile assessment by two independent examiners]
Time Frame: 3 years with assessment visits at baseline, 6 months, 1 year, 2 years, and 3 years
Population: as for outcome 1
Measure: Count of Units; unit: Restorations
Units Other Than Participants: Restorations
Arm/Group | CAD/CAM Onlays | CAD/CAM Crowns
Number analyzed (Participants) | 35 | 33
Number analyzed (Restorations) | 40 | 40
Restorations
  Baseline: 1: Clinically excellent | 40 | 40
  Baseline: 2: Clinically good | 0 | 0
  Baseline: Missed visit / no data | 0 | 0
  Baseline: Failed onlay / crown | 0 | 0
  6 months post-restoration: 1: Clinically excellent | 40 | 40
  6 months post-restoration: 2: Clinically good | 0 | 0
  6 months post-restoration: Missed visit / no data | 0 | 0
  6 months post-restoration: Failed onlay / crown | 0 | 0
  1 year post-restoration: 1: Clinically excellent | 39 | 39
  1 year post-restoration: 2: Clinically good | 0 | 0
  1 year post-restoration: Missed visit / no data | 1 | 1
  1 year post-restoration: Failed onlay / crown | 0 | 0
  2 years post-restoration: 1: Clinically excellent | 39 | 40
  2 years post-restoration: 2: Clinically good | 0 | 0
  2 years post-restoration: Missed visit / no data | 0 | 0
  2 years post-restoration: Failed onlay / crown | 1 | 0
  3 years post-restoration: 1: Clinically excellent | 38 | 39
  3 years post-restoration: 2: Clinically good | 0 | 0
  3 years post-restoration: Missed visit / no data | 1 | 1
  3 years post-restoration: Failed onlay / crown | 1 | 0

15. Secondary Outcome: Biologic Properties of Restorations (Onlays and Crowns) [Post-operative Sensitivity]
Description: Post-operative sensitivity. Evaluations according to FDI World Dental Federation criteria (Hickel et al., 2010) [1: Clinically excellent, 2: Clinically good, 3: Clinically sufficient, 4: Clinically unsatisfactory, 5: Clinically poor] Biological properties assessed by patient interview.]
Time Frame: 3 years with assessments at 6 months, 1 year, 2 years, and 3 years
Population: as for outcome 1
Measure: Count of Units; unit: Restorations
Units Other Than Participants: Restorations
Arm/Group | CAD/CAM Onlays | CAD/CAM Crowns
Number analyzed (Participants) | 35 | 33
Number analyzed (Restorations) | 40 | 40
Restorations
  6 months post-restoration: 1: Clinically excellent | 40 | 39
  6 months post-restoration: 2: Clinically good | 0 | 1
  6 months post-restoration: Missed visit / no data | 0 | 0
  6 months post-restoration: Failed onlay / crown | 0 | 0
  1 year post-restoration: 1: Clinically excellent | 39 | 37
  1 year post-restoration: 2: Clinically good | 0 | 2
  1 year post-restoration: Missed visit / no data | 1 | 1
  1 year post-restoration: Failed onlay / crown | 0 | 0
  2 years post-restoration: 1: Clinically excellent | 39 | 40
  2 years post-restoration: 2: Clinically good | 0 | 0
  2 years post-restoration: Missed visit / no data | 0 | 0
  2 years post-restoration: Failed onlay / crown | 1 | 0
  3 years post-restoration: 1: Clinically excellent | 38 | 39
  3 years post-restoration: 2: Clinically good | 0 | 0
  3 years post-restoration: Missed visit / no data | 1 | 1
  3 years post-restoration: Failed onlay / crown | 1 | 0

16. Secondary Outcome: Esthetic Properties of Restorations (Onlays and Crowns) [Surface Staining Scores]
Description: Surface Staining: Evaluations according to FDI World Dental Federation criteria (Hickel et al., 2010) [1: Clinically excellent, 2: Clinically good, 3: Clinically sufficient, 4: Clinically unsatisfactory, 5: Clinically poor]
Time Frame: 3 years with assessment visits at baseline, 6 months, 1 year, 2 years, and 3 years
Population: as for outcome 1
Measure: Count of Units; unit: Restorations
Units Other Than Participants: Restorations
Arm/Group | CAD/CAM Onlays | CAD/CAM Crowns
Number analyzed (Participants) | 35 | 33
Number analyzed (Restorations) | 40 | 40
Restorations
  Baseline: 1: Clinically excellent | 40 | 40
  Baseline: 2: Clinically good | 0 | 0
  Baseline: Missed visit, no data | 0 | 0
  Baseline: Failed onlay / crown | 0 | 0
  6 months post-restoration: 1: Clinically excellent | 40 | 40
  6 months post-restoration: 2: Clinically good | 0 | 0
  6 months post-restoration: Missed visit, no data | 0 | 0
  6 months post-restoration: Failed onlay / crown | 0 | 0
  1 year post-restoration: 1: Clinically excellent | 39 | 39
  1 year post-restoration: 2: Clinically good | 0 | 0
  1 year post-restoration: Missed visit, no data | 1 | 1
  1 year post-restoration: Failed onlay / crown | 0 | 0
  2 years post-restoration: 1: Clinically excellent | 39 | 40
  2 years post-restoration: 2: Clinically good | 0 | 0
  2 years post-restoration: Missed visit, no data | 0 | 0
  2 years post-restoration: Failed onlay / crown | 1 | 0
  3 years post-restoration: 1: Clinically excellent | 38 | 39
  3 years post-restoration: 2: Clinically good | 0 | 0
  3 years post-restoration: Missed visit, no data | 1 | 1
  3 years post-restoration: Failed onlay / crown | 1 | 0

17. Secondary Outcome: Esthetic Properties of Restorations (Onlays and Crowns) [Margin Staining Scores]
Description: Margin Staining: Evaluations according to FDI World Dental Federation criteria (Hickel et al., 2010) [1: Clinically excellent, 2: Clinically good, 3: Clinically sufficient, 4: Clinically unsatisfactory, 5: Clinically poor]
Time Frame: 3 years with assessment visits at baseline, 6 months, 1 year, 2 years, and 3 years
Population: as for outcome 1
Measure: Count of Units; unit: Restorations
Units Other Than Participants: Restorations
Arm/Group | CAD/CAM Onlays | CAD/CAM Crowns
Number analyzed (Participants) | 35 | 33
Number analyzed (Restorations) | 40 | 40
Restorations
  Baseline: 1: Clinically excellent | 40 | 40
  Baseline: 2: Clinically good | 0 | 0
  Baseline: Missed visit, no data | 0 | 0
  Baseline: Failed onlay / crown | 0 | 0
  6 months post-restoration: 1: Clinically excellent | 40 | 40
  6 months post-restoration: 2: Clinically good | 0 | 0
  6 months post-restoration: Missed visit, no data | 0 | 0
  6 months post-restoration: Failed onlay / crown | 0 | 0
  1 year post-restoration: 1: Clinically excellent | 39 | 39
  1 year post-restoration: 2: Clinically good | 0 | 0
  1 year post-restoration: Missed visit, no data | 1 | 1
  1 year post-restoration: Failed onlay / crown | 0 | 0
  2 years post-restoration: 1: Clinically excellent | 39 | 40
  2 years post-restoration: 2: Clinically good | 0 | 0
  2 years post-restoration: Missed visit, no data | 0 | 0
  2 years post-restoration: Failed onlay / crown | 1 | 0
  3 years post-restoration: 1: Clinically excellent | 38 | 39
  3 years post-restoration: 2: Clinically good | 0 | 0
  3 years post-restoration: Missed visit, no data | 1 | 1
  3 years post-restoration: Failed onlay / crown | 1 | 0

18. Secondary Outcome: Esthetic Properties of Restorations (Onlays and Crowns) [Color Match and Translucency Scores]
Description: Color Match and Translucency: Evaluations according to FDI World Dental Federation criteria (Hickel et al., 2010) [1: Clinically excellent, 2: Clinically good, 3: Clinically sufficient, 4: Clinically unsatisfactory, 5: Clinically poor]
Time Frame: 3 years with assessment visits at baseline, 6 months, 1 year, 2 years, and 3 years
Population: as for outcome 1
Measure: Count of Units; unit: Restorations
Units Other Than Participants: Restorations
Arm/Group | CAD/CAM Onlays | CAD/CAM Crowns
Number analyzed (Participants) | 35 | 33
Number analyzed (Restorations) | 40 | 40
Restorations
  Baseline: 1: Clinically excellent | 40 | 40
  Baseline: 2: Clinically good | 0 | 0
  Baseline: Missed visit, no data | 0 | 0
  Baseline: Failed onlay / crown | 0 | 0
  6 months post-restoration: 1: Clinically excellent | 39 | 40
  6 months post-restoration: 2: Clinically good | 1 | 0
  6 months post-restoration: Missed visit, no data | 0 | 0
  6 months post-restoration: Failed onlay / crown | 0 | 0
  1 year post-restoration: 1: Clinically excellent | 39 | 39
  1 year post-restoration: 2: Clinically good | 0 | 0
  1 year post-restoration: Missed visit, no data | 1 | 1
  1 year post-restoration: Failed onlay / crown | 0 | 0
  2 years post-restoration: 1: Clinically excellent | 39 | 40
  2 years post-restoration: 2: Clinically good | 0 | 0
  2 years post-restoration: Missed visit, no data | 0 | 0
  2 years post-restoration: Failed onlay / crown | 1 | 0
  3 years post-restoration: 1: Clinically excellent | 38 | 39
  3 years post-restoration: 2: Clinically good | 0 | 0
  3 years post-restoration: Missed visit, no data | 1 | 1
  3 years post-restoration: Failed onlay / crown | 1 | 0

19. Secondary Outcome: Esthetic Properties of Restorations (Onlays and Crowns) [Aesthetic Anatomical Form Scores]
Description: Aesthetic anatomical form: Evaluations according to FDI World Dental Federation criteria (Hickel et al., 2010) [1: Clinically excellent, 2: Clinically good, 3: Clinically sufficient, 4: Clinically unsatisfactory, 5: Clinically poor]
Time Frame: 3 years with assessment visits at baseline, 6 months, 1 year, 2 years, and 3 years
Population: as for outcome 1
Measure: Count of Units; unit: Restorations
Units Other Than Participants: Restorations
Arm/Group | CAD/CAM Onlays | CAD/CAM Crowns
Number analyzed (Participants) | 35 | 33
Number analyzed (Restorations) | 40 | 40
Restorations
  Baseline: 1: Clinically excellent | 40 | 40
  Baseline: 2: Clinically good | 0 | 0
  Baseline: Missed visit, no data | 0 | 0
  Baseline: Failed onlay / crown | 0 | 0
  6 months post-restoration: 1: Clinically excellent | 40 | 40
  6 months post-restoration: 2: Clinically good | 0 | 0
  6 months post-restoration: Missed visit, no data | 0 | 0
  6 months post-restoration: Failed onlay / crown | 0 | 0
  1 year post-restoration: 1: Clinically excellent | 39 | 39
  1 year post-restoration: 2: Clinically good | 0 | 0
  1 year post-restoration: Missed visit, no data | 1 | 1
  1 year post-restoration: Failed onlay / crown | 0 | 0
  2 years post-restoration: 1: Clinically excellent | 39 | 40
  2 years post-restoration: 2: Clinically good | 0 | 0
  2 years post-restoration: Missed visit, no data | 0 | 0
  2 years post-restoration: Failed onlay / crown | 1 | 0
  3 years post-restoration: 1: Clinically excellent | 38 | 39
  3 years post-restoration: 2: Clinically good | 0 | 0
  3 years post-restoration: Missed visit, no data | 1 | 1
  3 years post-restoration: Failed onlay / crown | 1 | 0

ADVERSE EVENTS:
Time Frame: From participant's first treatment restoration to subject's completion of the study, an average of 3 years..
Description: Non-device related adverse event reporting was not required beyond the 6-month follow-up visit. Reporting of all device-related and serious adverse events was required throughout the study (3 years).
Arm/Group | CAD/CAM Onlays | CAD/CAM Crowns
All-Cause Mortality (participants affected / at risk) | 1/35 | 0/33
Serious Adverse Events (participants affected / at risk) | 1/35 | 0/33
Other Adverse Events (participants affected / at risk) | 0/35 | 0/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CAD/CAM Onlays (N=35) | CAD/CAM Crowns (N=33)
Death (General disorders) | 1 (1) | 0 (0) — Non-device related. Patient records are locked, not available to dental clinic. No other information is available. Cause and date unknown.

LIMITATIONS AND CAVEATS:
Assessments were planned to be examined by two independent clinical evaluators using pre-defined Fédération Dentaire Internationale (FDI) criteria. However, some of the evaluations were made by only a single evaluator. Each occurrence was recorded in the study file as a protocol deviation and was not expected to affect the conclusions of the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-02-17): https://cdn.clinicaltrials.gov/large-docs/74/NCT04279574/Prot_SAP_000.pdf